CLINICAL TRIAL: NCT04589650
Title: EPIK-P2: A Phase II Double-blind Study With an Upfront, 16-week Randomized, Placebo-controlled Period, to Assess the Efficacy, Safety and Pharmacokinetics of Alpelisib (BYL719) in Pediatric and Adult Patients With PIK3CA-related Overgrowth Spectrum (PROS)
Brief Title: Study Assessing the Efficacy, Safety and PK of Alpelisib (BYL719) in Pediatric and Adult Patients With PIK3CA-related Overgrowth Spectrum
Acronym: EPIK-P2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBYL719F12201; 2023-508530-34-00 (Registry Identifier: EU CT Number)
Expanded Access: NCT04085653 (Available)
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: PIK3CA-related Overgrowth Spectrum (PROS)
Keywords: PIK3CA-related overgrowth spectrum (PROS); Alpelisib; BYL719; Adult; Pediatric; Phase II
MeSH Terms: interventions — Alpelisib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigator staff, and persons performing the assessments will remain blinded to the identity of the treatment from the time of randomization until primary analysis i.e. the last participants (Groups 1 and 2) completes Week 48 from randomization or discontinues earlier.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Adult cohort (group 1)- Alpelisib (Experimental): During double-blind randomized study period (from baseline up to Week 16), adult participants will be randomized to receive alpelisib (125 mg, oral, once daily). After Week 16, participants will continue their active treatment at the same dose level.
  Interventions: Drug: Alpelisib
- Adult cohort (group 1)- Placebo (Placebo Comparator): During double-blind randomized study period (from baseline up to Week 16), adult participants will be randomized to receive placebo. After Week 16, participants will be switched to active treatment with alpelisib at the placebo dose level received at the end of the placebo period.
  Interventions: Drug: Alpelisib; Drug: Placebo
- Pediatric cohort (group 2: 6 to 17 years old) -Alpelisib (Experimental): During double-blind randomized study period (from baseline up to Week 16, pediatric participants (6 to 17 years old) will be randomized to receive alpelisib (50 mg, oral, once daily). After Week 16, participants will continue their active treatment at the same dose level.
  Interventions: Drug: Alpelisib
- Pediatric cohort (group 2: 6 to 17 years old)-Placebo (Placebo Comparator): During double-blind randomized study period (from baseline up to Week 16), pediatric participants (6 to 17 years old) will be randomized to receive Placebo. After Week 16, participants will be switched to active treatment with alpelisib at the placebo dose level received at the end of the placebo period.
  Interventions: Drug: Alpelisib; Drug: Placebo
- Pediatric cohort (group 3: 0 to 5 years old)- Alpelisib granules (Experimental): Pediatric participants (0 to 5 years old) will receive alpelisib granules formulation with an age-dependent starting dose (<1 month: 20 mg every other day; 1 to <6 months: 20 mg daily; 6 to <2 years: 40 mg daily; 2 to <6 years: 50 mg daily).
  Interventions: Drug: Alpelisib
- Pediatric cohort (group 4: 2 to 5 years old)- Alpelisib FCT (Experimental): Pediatric participants (2 to 5 years old) will receive 50 mg of alpelisib film-coated tablets (FCT) once daily in an open-label setting.
  Interventions: Drug: Alpelisib
- Pediatric cohort (group 5: 6-17 years old)-Alpelisib FCT (Experimental): Pediatric participants (6 to 17 year old) will receive 125 mg alpelisib film-coated (FCT) once daily, in an open-label setting.
  Interventions: Drug: Alpelisib

INTERVENTIONS:
Drug: Alpelisib — Adult participants (group 1) will receive 125 mg of alpelisib oral tablets once daily. Pediatric participants (Group 2: 6 to 17 years old) will receive 50 mg of alpelisib oral tablets once daily. Pediatric participants (Group 4: 2 to 5 years old) will receive 50 mg of alpelisib oral tablets once daily, Pediatric participants (Group 3: 0 to 5 years old) will receive alpelisib granules formulation with an age-dependent starting dose and maximum dose levels ranging from 20 mg every other day to 50 mg once daily. Pediatric participants (Group 5: 6 to 17 years old) will receive 125 mg of alpelisib oral tablets once daily.
  Other Names: BYL719
Drug: Placebo — Participants will receive matching placebo once daily up to week 16.
  Arms: Adult cohort (group 1)- Placebo; Pediatric cohort (group 2: 6 to 17 years old)-Placebo

SUMMARY:
This is a prospective Phase II multi-center study with an initial 16-week, randomized, double-blind, placebo-controlled period, followed by two extension periods to assess the efficacy, safety and pharmacokinetics (PK) of alpelisib in pediatric and adult patients with PIK3CA-related overgrowth spectrum (PROS)

DETAILED DESCRIPTION:
This is a Phase II multi-center study with an upfront 16-week, randomized, double-blind, placebo-controlled period, and extension periods, to assess the efficacy, safety and PK of alpelisib in pediatric and adult participants with PROS.

Study period 1 - Core Period: Double-blind treatment, with an upfront 16-week placebo-controlled period (From Randomization to the end of Week 24) - Groups 1 and 2 At study start, participants in Group 1 and Group 2 will be enrolled and randomized in a 2:1 ratio (104 participants in the active arms and 52 participants in the placebo arms) to alpelisib or matching placebo. The upfront placebo-controlled period will continue for the first 16 weeks. At the conclusion of week 16, those participants who were randomized to receive placebo will be switched to active treatment with alpelisib in a blinded fashion at the dose level received at the end of the placebo period. Those participants who were randomized to receive alpelisib, will continue their treatment at the same dose level.

During the initial 16 weeks of the Core period, study treatment will be given in a blinded fashion, starting from week 17 of the Core period in open label fashion. The randomized treatment assignment to the treatment arms will remain blinded to participants, Investigators and the study team until the time of the primary analysis, when the last participant reaches week 48 from randomization or discontinues earlier.

Study period 1 - Exploratory; Group 4, open label treatment with the alpelisib FCT formulation After the implementation of Global Protocol Amendment 01, approximately 6 participants 2 to 5 years of age will be enrolled in exploratory Group 4. These participants will receive alpelisib FCT in an open label setting.

Study period 2 - Extension 1: treatment with alpelisib (week 25 up to the end of week 48) - Groups 1 and 2 Participants (Group 1 and Group 2) will continue their treatment during this study period.

For Groups 1 and 2, dose escalation is NOT allowed during first 4 weeks of Extension 1 period (weeks 25-28).

Once a participant (Groups 1 and 2) has completed initial 24 weeks of study treatment and reached Week 29, dose escalation will be allowed (Refer to Section 6.5.1):

* Group 1: Alpelisib (125mg, or 200mg, or 250 mg QD)
* Group 2: Alpelisib (50mg, or 125mg, or 200mg, or 250 mg QD)

Study period 2 - Exploratory: Group 4, open label treatment with the alpelisib FCT formulation

For Group 4 dose escalation is allowed once participant has reached the age of 6 years old, has completed the initial 24 weeks of study treatment, and has reached week 25:

• Group 4: Alpelisib (50 mg, or 125 mg, or 200 mg, or 250 mg QD)

Study period 3 - Extension 2: long-term treatment with alpelisib (Week 49 up to 5 years) - Groups 1 and 2 Groups 1 and 2 participants who continue the study until Week 48 and have clinical benefit from the study treatment, will enter a long-term extension period. Dose escalation and treatment beyond progression are allowed in both Group 1 and Group 2.

Study period 3 - Exploratory: Group 4, open label treatment with the alpelisib FCT formulation Group 4 participants who continue the study until Week 48 and have clinical benefit from the study treatment, will enter a long-term extension period. Dose escalation is allowed once a participant has reached the age of 6 years old, has completed the initial 24 weeks of study treatment, and has reached Week 25.

Exploratory study part: Group 3, open label treatment with the alpelisib granules formulation Group 3 will be an exploratory group of participants who are 0 to 5 years old and will receive the alpelisib granules formulation with an age-dependent starting dose and maximum dose levels ranging from 20 mg every other day to 50 mg once daily. Group 3 will be open to enrollment only after implementation of Global Protocol Amendment 05. Dose escalation is allowed once a participant has reached the age of 6 years, has completed the initial 24 weeks of study treatment, and has reached Week 25.

Group 5 open-label treatment with the alpelisib FCT formulation:

Participants of Group 5 will be enrolled after implementation of Global Protocol Amendment 02 and immediately after enrollment of Group 2 has been completed and will receive a starting dose of 125 mg alpelisib FCT formulation once daily in an open-label setting.

Dose escalation is allowed for those who did not derive sufficient clinical benefit at the Investigator's discretion and once participant has reached at least Week 25.

Study period 4 - Extension 3: treatment with alpelisib (from Week 264 until last patient enrolled completes 5 years of treatment) All participants from all groups will be followed until the last patient enrolled completes 5 years of treatment or discontinues early, to collect additional safety of alpelisib and in order to ensure patient access to treatment in the absence of global commercial supply in pediatric and adult participants with PROS. Visits will be performed every 24 weeks and additional safety assessments every 48 weeks.

It is planned to enroll approximately 192 participants in total, 78 adults and 114 children and adolescents. A total of approximately 156 male or female participants (of age ≥ 6 years) with PROS will be randomized in a 2:1 ratio in Groups 1 and 2 (approximately 78 participants per age group). Additional exploratory groups (Group 3, Group 4 and Group 5) will include approximately a total of 36 participants (approximately 15 in Group 3, 6 in Group 4 and 15 in Group 5).

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent and assent (when applicable) from the patient, parent, legal authorized representative, or guardian prior to any study-related screening procedures were performed.
* Male or female patients age above 0 day at the time of informed consent: Group 1: ≥ 18 years old, Group 2: 6-17 years old, Group 3: ≥ 0-5 years old, Group 4: ≥ 2-5 years old, Group 5: 6-17 years old.
* Patients with diagnosis of PROS with symptomatic and /or progressive overgrowth and at least one measurable PROS-related lesion confirmed by BIRC assessment who had syndromic disease or isolated features at the time of informed consent. Patients, who previously had been receiving systemic treatment for PROS, could enter the study.
* Documented evidence of a somatic mutation(s) in the PIK3CA gene performed in local laboratories using a DNA-based test validated according to the local regulations at the time of informed consent.
* A tissue sample (fresh or archival) was to be sent to a Novartis-designated central laboratory.
* Karnofsky (in patients > 16 years old at study entry)/Lansky (≤ 16 years of age at study entry) performance status index ≥ 50.
* Adequate bone marrow and organ function as assessed by central laboratory for eligibility.
* Presence of at least one PROS-related measurable lesion defined as a lesion with longest diameter ≥ 2 cm, when the volume could be accurately and reproducibly measured by MRI, and associated with complaints, clinical symptoms or functional limitations affecting the patient's everyday life. Measurability was confirmed by BIRC before randomization.
* Able to swallow study drug (as assessed within 7 days before study treatment start):
* Groups 1, 2, 4, and 5: FCT, or as drinkable suspension when applicable.
* Group 3: granules. Drug administration via feeding tube is allowed.

Key Exclusion Criteria:

* Patient with only isolated macrodactyly, epidermal nevus/nevi and macroencephaly (the only clinical feature or a combination of any three of them), in absence of other PROS-related lesions at the time of informed consent.
* Previous treatment with alpelisib and/or any other PI3K inhibitor(s).
* Radiation exposure for PROS treatment purpose within the previous 12 months on those PROS areas, which were expected to qualify for target lesions (except lesion(s) progressing after completion of radiotherapy) at time of informed consent.
* Debulking or other major surgery performed within 3 months at time of informed consent.
* Clinically meaningful bleeding related to PROS: Grade 2 within 14 days or grade 3 and more within 28 days before study treatment start as per CTCAE v4.03.
* Clinically meaningful PROS-related thrombotic event (grade 2 and more as per CTCAE v4.03) within 30 days before informed consent, and/or sclerotherapy/embolization for vascular complications performed within 6 weeks before informed consent.
* History of prior and or ongoing malignancy or ongoing investigations or treatment for malignancy at time of informed consent.
* Clinically significant heart disease at time of informed consent.
* Patients in Groups 1, 2, and 5 with documented pneumonitis or interstitial lung disease at time of informed consent and with impaired lung function (e.g., FEV1 or DLCO ≤ 70% of predicted) that was not related to PROS. Patients in Groups 3 and 4 with documented or suspicious pneumonitis or interstitial lung disease based on MRI images at time of informed consent.
* History of acute pancreatitis within 1 year before informed consent or past medical history of chronic pancreatitis at time of informed consent.
* Patients with an established diagnosis of type I diabetes mellitus or uncontrolled type II diabetes mellitus at time of informed consent.
* Known impairment of gastrointestinal (GI) function due to concomitant GI disease that may significantly alter the absorption of the study drug at time of informed consent.
* History of hypersensitivity to any drugs or metabolites of PI3K inhibitor or any of the excipients of alpelisib at time of informed consent.
* Known history of Steven Johnson's syndrome, erythema multiforme or toxic epidermal necrolysis at time of informed consent.
* Known history of seizure, or epilepsy, regardless of relatedness to PROS spectrum at time of informed consent, when epilepsy was not controlled and/or the patient may not be switched to non-enzyme inducing antiepileptic drug(s) at time of informed consent.
* Patient with other concurrent severe and/or uncontrolled medical conditions that could, in the Treating Physician's judgment, contraindicate administration of alpelisib at time of informed consent. Patient with an active documented COVID-19 infection at time of informed consent could be included only when completely recovered and had no symptoms for at least 28 days before first dose of study medication.
* Pregnant or breastfeeding female patients at time of informed consent.
* Female patients of child-bearing potential who did not consent to use a highly effective method of contraception and male patients who did not consent to use a condom and/or a highly effective method of contraception for the duration of the study and for one week following discontinuation of alpelisib.
* Patient was receiving any of the following medications and could not discontinue 7 days prior to the start of the treatment: strong inducers of CYP3A4 or inhibitors of breast cancer resistance protein (BCRP).
* Not able to understand and to comply with study instructions and requirements at time of informed consent.
* Participation in a prior investigational study within 4 weeks prior to study treatment start or within 5 half-lives of the investigational product, whichever was longer.
* Patients with clinically significant worsening of PROS-related laboratory anomalies, physical signs and symptoms indicating an uncontrolled condition during the screening phase, particularly if systemic treatment with any other inhibitor of the PI3K/AKT/mTOR pathway was stopped prior to the start of study treatment. This included but was not limited to hypercoagulability state in patients not receiving prophylactic treatment.

Other inclusion/exclusion criteria may apply

Ages: 0 Days to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2031-01-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- United States (11):
  - UCSF Birthmarks and Vascular Center, San Francisco, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Washington Univ School Of Medicine, St Louis, Missouri
  - Fink Childrens Ambulatory Care Ctr, New York, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children s Hospital Medical Center, Cincinnati, Ohio
  - Cinn Children Hosp Medical Center, Cincinnati, Ohio
  - CHOP Abramson Pediatric Resch Ctr, Philadelphia, Pennsylvania
  - Unv of TX Southwestern Medical Center, Dallas, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Childrens Hospital and Regional Medical Center, Seattle, Washington
- Novartis Investigative Site, Montreal, Quebec, Canada
- China (2):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- France (4):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Tours
- Germany (5):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
- Novartis Investigative Site, Pokfulam, Hong Kong
- Italy (2):
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
- Novartis Investigative Site, Nijmegen, Gelderland, Netherlands
- Novartis Investigative Site, Oslo, Norway
- Spain (2):
  - Novartis Investigative Site, Esplugues, Barcelona
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Zurich
- United Kingdom (3):
  - Novartis Investigative Site, West Midlands, Birmingham
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Fujino A, Kuniyeda K, Nozaki T, Ozeki M, Ohyama T, Sato I, Kamibeppu K, Tanaka A, Uemura N, Kanmuri K, Nakamura K, Kobayashi F, Suenobu S, Nomura T, Hayashi A, Nagao M, Kato A, Aramaki-Hattori N, Imagawa K, Ishikawa K, Ochi J, Horiuchi S, Nagabukuro H. The Prospective Natural History Study of Patients with Intractable Venous Malformation and Klippel-Trenaunay Syndrome to Guide Designing a Proof-of-Concept Clinical Trial for Novel Therapeutic Intervention. Lymphat Res Biol. 2024 Feb;22(1):27-36. doi: 10.1089/lrb.2023.0023. Epub 2023 Dec 19. PMID 38112724
- [Derived] Madsen RR, Semple RK. PIK3CA-related overgrowth: silver bullets from the cancer arsenal? Trends Mol Med. 2022 Apr;28(4):255-257. doi: 10.1016/j.molmed.2022.02.009. Epub 2022 Mar 8. PMID 35272946

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is conducted globally across 12 countries. Recruitment in Group 3 will be open after protocol amendment 5 approval in 2025.
Groups:
- Group 1 (Greater or Equal to 18 Years) - Alpelisib Arm: Group 1 (Greater or equal to 18 years): During double-blind randomized study period (from baseline up to Week 16), adult participants will be randomized to receive alpelisib (125 mg, oral, once daily). After Week 16, participants will continue their active treatment at the same dose level.
- Group 1 (Greater or Equal to 18 Years) - Placebo Arm: Group 1: During double-blind randomized study period (from baseline up to Week 16), adult participants will be randomized to receive placebo (125 mg, oral, once daily). After Week 16, participants will be switched to active treatment with alpelisib at the placebo dose level received at the end of the placebo period.
- Group 2 (6-17 Years) - Alpelisib Arm: Group 2: During double-blind randomized study period (from baseline up to Week 16, pediatric participants (6 to 17 years old) will be randomized to receive alpelisib (50 mg, oral, once daily). After Week 16, participants will continue their active treatment at the same dose level.
- Group 2 (6-17 Years) - Placebo Arm: Group 2: During double-blind randomized study period (from baseline up to Week 16), pediatric participants (6 to 17 years old) will be randomized to receive Placebo (50mg, oral, once daily). After Week 16, participants will be switched to active treatment with alpelisib at the placebo dose level received at the end of the placebo period.
- Exploratory Group 4 (2-5 Years) All Pediatrics - Alpelisib FCT: Pediatric participants (2 to 5 years old) will receive 50 mg of alpelisib film-coated tablets (FCT) once daily in an open-label setting.
- Exploratory Group 5 (6-17 Years) All Pediatrics - Alpelisib FCT: Pediatric participants (6 to 17 year old) will receive 125 mg alpelisib film-coated (FCT) once daily, in an open-label setting.
Period: Overall Study
Arm/Group | Group 1 (Greater or Equal to 18 Years) - Alpelisib Arm | Group 1 (Greater or Equal to 18 Years) - Placebo Arm | Group 2 (6-17 Years) - Alpelisib Arm | Group 2 (6-17 Years) - Placebo Arm | Exploratory Group 4 (2-5 Years) All Pediatrics - Alpelisib FCT | Exploratory Group 5 (6-17 Years) All Pediatrics - Alpelisib FCT
Started | 54 | 27 | 56 | 28 | 7 | 16
Completed Core (Patients who completed a study period (i.e., Core, Extension 1) are continuing into the next study period.) | 52 | 26 | 55 | 26 | 7 | 13
Completed Extension 1 (Patients who completed a study period (i.e., Core, Extension 1) are continuing into the next study period.) | 46 | 24 | 55 | 26 | 7 | 4
Full Analysis Set (FAS) (Groups 1 and 2 = all patients to whom study treatment was assigned by randomization. Groups 4 and 5 = all patients to whom study treatment had been assigned and who received at least one dose of study treatment.) | 54 (All patients to whom study treatment was assigned by randomization.) | 27 (All patients to whom study treatment was assigned by randomization.) | 56 (All patients to whom study treatment was assigned by randomization.) | 28 (All patients to whom study treatment was assigned by randomization.) | 7 (All patients to whom study treatment had been assigned and who received at least one dose of study treatment.) | 16 (All patients to whom study treatment had been assigned and who received at least one dose of study treatment.)
Full Analysis Set (FAS) - BYL719 (All patients to whom alpelisib had been assigned by randomization. This analysis set was used for the analysis of the primary endpoint.) | 54 | 0 | 56 | 0 | 0 | 0
Safety Set (All patients who received at least one dose of study treatment) | 54 | 27 | 56 | 28 | 7 | 16
Pharmacokinetic Analysis Set (PAS) (All patients who received at least one dose of alpelisib and provided at least one evaluable PK concentration.) | 51 | 25 | 56 | 26 | 7 | 16
Completed (Started - Discontinued at anytime) | 42 | 23 | 53 | 25 | 7 | 15
Not Completed | 12 | 4 | 3 | 3 | 0 | 1
Not completed — Subject decision | 6 | 2 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 1 | 1 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Guardian Decision | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Greater or Equal to 18 Years) - Alpelisib Arm | Group 1 (Greater or Equal to 18 Years) - Placebo Arm | Group 2 (6-17 Years) - Alpelisib Arm | Group 2 (6-17 Years) - Placebo Arm | Exploratory Group 4 (2-5 Years) All Pediatrics - Alpelisib FCT | Exploratory Group 5 (6-17 Years) All Pediatrics - Alpelisib FCT | Total
Number analyzed (Participants) | 54 | 27 | 56 | 28 | 7 | 16 | 188
Age, Customized [Count of Participants; unit: Participants]
  Children, 2 - < 6 years | 0 | 0 | 0 | 0 | 7 | 0 | 7
  Children, 6 - < 12 years | 0 | 0 | 28 | 19 | 0 | 12 | 59
  Adolescent, 12 - < 18 years | 0 | 0 | 28 | 9 | 0 | 4 | 41
  18 - < 65 years | 54 | 27 | 0 | 0 | 0 | 0 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 14 | 27 | 12 | 3 | 8 | 98
  Male | 20 | 13 | 29 | 16 | 4 | 8 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 3 | 10 | 3 | 0 | 2 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 0 | 0 | 2
  White | 48 | 22 | 42 | 25 | 7 | 13 | 157
  More than one race | 0 | 1 | 2 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Randomized to Alpelisib With a Confirmed Objective Response by BIRC in Group 1 and Group 2
Description: A responder is defined by achieving a >=20% reduction from baseline in the sum of target lesion volumes (via BIRC), provided that none of the individual target lesions have a >=20% increase from baseline and in absence of progression of non target lesions and without new lesions. Confirmation of response requires a subsequent imaging assessment performed at least 4 weeks after the onset of response. Participants who permanently discontinued alpelisib prior to confirmation of response, and participants who received surgery as rescue therapy prior to confirmation of response are considered as non-responders.
Time Frame: Up to 48 weeks
Population: Full Analysis Set (FAS) - BYL719. All patients to whom alpelisib had been assigned by randomization.
Measure: Number (97.5% Confidence Interval); unit: % of confirmed responder by BIRC
Arm/Group | Group 1 (Greater or Equal to 18 Years) - Alpelisib Arm | Group 2 (6-17 Years) - Alpelisib Arm
Number analyzed (Participants) | 54 | 56
% of confirmed responder by BIRC | 16.7 [7.0 to 31.1] | 23.2 [11.9 to 38.3]

2. Secondary Outcome: Key Secondary Objective: Proportion of Participants With Response at Week 16 by BIRC in Group 1 and Group 2
Description: A responder is defined by achieving a >=20% reduction from baseline in the sum of target lesion volumes (via BIRC) at Week 16, provided that none of the individual target lesions have a >=20% increase from baseline and in absence of progression of non-target lesions and without new lesions. Participants who permanently discontinued alpelisib prior to Week 16, participants who received surgery as rescue therapy prior to Week 16, and participants who had a missing/non-evaluable radiological assessment at Week 16 are considered as non-responders.
Time Frame: Week 16
Population: Full Analysis Set (FAS). All patients to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: % of responder by BIRC
Arm/Group | Group 1 (Greater or Equal to 18 Years) - Alpelisib Arm | Group 1 (Greater or Equal to 18 Years) - Placebo Arm | Group 2 (6-17 Years) - Alpelisib Arm | Group 2 (6-17 Years) - Placebo Arm
Number analyzed (Participants) | 54 | 27 | 56 | 28
% of responder by BIRC | 11.1 [4.2 to 22.6] | 0 [0.0 to 12.8] | 8.9 [3.0 to 19.6] | 0 [0.0 to 12.3]

3. Secondary Outcome: Proportion of Participants With a Response at Week 24 (by BIRC) in Groups 1 and 2
Description: A responder is defined by achieving a >=20% reduction from baseline in the sum of target lesion volumes (via BIRC) at Week 24, provided that none of the individual target lesions have a >=20% increase from baseline and in absence of progression of non-target lesions and without new lesions.
Time Frame: Week 24
Population: Full Analysis Set (FAS) - BYL719. All patients to whom alpelisib had been assigned by randomization.
Measure: Number (97.5% Confidence Interval); unit: % of confirmed responder by BIRC
Arm/Group | Group 1 (Greater or Equal to 18 Years) - Alpelisib Arm | Group 2 (6-17 Years) - Alpelisib Arm
Number analyzed (Participants) | 54 | 56
% of confirmed responder by BIRC | 16.7 [7 to 31.1] | 19.6 [9.2 to 34.3]

4. Secondary Outcome: Frequency and Severity of Adverse Events in Groups 1 and 2 up to Week 16
Description: An adverse event (AE) is any untoward medical occurrence (e.g., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a participant or clinical investigation participant after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product. This includes events reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative).
  Treatment emergent Adverse Event (TEAEs) in this study are events that started after the first dose of study treatment and until 30 days after the last dose of study treatment, or events present prior to the first dose of treatment which increased in severity based on preferred term within 30 days after the last study treatment.
Time Frame: Up to Week 16
Population: Safety Set. All patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Greater or Equal to 18 Years) - Alpelisib Arm | Group 1 (Greater or Equal to 18 Years) - Placebo Arm | Group 2 (6-17 Years) - Alpelisib Arm | Group 2 (6-17 Years) - Placebo Arm
Number analyzed (Participants) | 54 | 27 | 56 | 28
Participants
  Adverse Events (AEs) | 50 | 26 | 50 | 24
  Treatment-related AEs | 31 | 12 | 19 | 9
  AEs with grade >=3 | 11 | 5 | 7 | 2
  Treatment-related AEs with grade >=3 | 5 | 1 | 3 | 0
  Serious Adverse Events (SAEs) | 5 | 2 | 3 | 2
  Treatment-related SAEs | 3 | 0 | 1 | 0
  AEs leading to discontinuation | 1 | 0 | 0 | 0
  Treatment-related AEs leading to discontinuation | 1 | 0 | 0 | 0
  AEs leading to dose adjustment/interruption | 6 | 6 | 4 | 4
  AEs leading to dose reduction | 0 | 0 | 0 | 0
  AEs leading to dose interruption | 6 | 6 | 4 | 4
  AEs requiring additional therapy | 37 | 19 | 43 | 15

5. Secondary Outcome: Frequency and Severity of Adverse Events in All Groups of Participants Over Time
Description: Type, frequency, seriousness, and severity of treatment-emergent adverse events per CTCAE v4.03 criteria in participants with PROS over time.
Time Frame: Up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2032-04

6. Secondary Outcome: Change From Baseline to Week 16 in Brief Pain Inventory (BPI) Worst Pain Intensity in Group 1 and 2
Description: For adult and pediatric patients 12 years of age and older, the BPI item that assesses worst pain intensity in the past 24 hours was used. Patients respond to the item on an 11-point response scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine). Worst pain intensity was averaged weekly over a 7-day period if a patient had completed the questionnaire for at least 4 days in the 7-day period. The weekly mean was calculated based on the available assessments. Clinically important change at Week 16 was defined as a 2-point reduction for patients who had a pain intensity score ≥ 4 at baseline. For patients with a baseline score < 4, a 1-point reduction from baseline was also considered as a clinically important change.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: Full Analysis Set (FAS). Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group 1 (Greater or Equal to 18 Years) - Alpelisib Arm | Group 1 (Greater or Equal to 18 Years) - Placebo Arm | Group 2 (6-17 Years) - Alpelisib Arm | Group 2 (6-17 Years) - Placebo Arm
Number analyzed (Participants) | 34 | 13 | 16 | 5
Score on a scale
  Change from BL at Week 4: number analyzed (Participants) | 30 | 10 | 14 | 4
  Change from BL at Week 4 | -0.9 (1.87) | -0.2 (1.54) | 0.2 (0.73) | 0.3 (0.82)
  Change from BL at Week 8: number analyzed (Participants) | 29 | 9 | 13 | 5
  Change from BL at Week 8 | -1.2 (2.13) | -0.7 (1.43) | -0.3 (0.91) | 0.1 (0.69)
  Change from BL at Week 12: number analyzed (Participants) | 27 | 8 | 13 | 4
  Change from BL at Week 12 | -0.9 (2.55) | -0.8 (1.41) | -0.4 (1.01) | 0.4 (0.62)
  Change from BL at Week 16: number analyzed (Participants) | 24 | 7 | 10 | 3
  Change from BL at Week 16 | -1.3 (2.46) | -0.1 (1.49) | -0.4 (1.34) | 0.3 (1.14)

7. Secondary Outcome: Number of Participants With Global Impression of Symptom Severity (PGIS) Score up to Week 16
Description: A Patient Global Impression of Symptom Severity item was used to understand the overall severity of symptoms experienced and clinical meaningfulness of treatment effects experienced during this study. This item included 5 response options: no symptoms, mild, moderate, severe, and very severe.
Time Frame: Week 4, Week 8, Week 16
Population: Full Analysis Set (FAS). Only participants with an available value for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Greater or Equal to 18 Years) - Alpelisib Arm | Group 1 (Greater or Equal to 18 Years) - Placebo Arm | Group 2 (6-17 Years) - Alpelisib Arm | Group 2 (6-17 Years) - Placebo Arm
Number analyzed (Participants) | 53 | 26 | 28 | 8
Participants
  Week 4: number analyzed (Participants) | 53 | 26 | 25 | 8
  Week 4: No symptoms | 12 | 9 | 15 | 3
  Week 4: Mild | 20 | 5 | 6 | 3
  Week 4: Moderate | 14 | 10 | 4 | 2
  Week 4: Severe | 6 | 2 | 0 | 0
  Week 4: Very severe | 1 | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 50 | 26 | 28 | 8
  Week 8: No symptoms | 12 | 7 | 17 | 3
  Week 8: Mild | 20 | 6 | 6 | 2
  Week 8: Moderate | 11 | 10 | 4 | 3
  Week 8: Severe | 7 | 1 | 1 | 0
  Week 8: Very severe | 0 | 2 | 0 | 0
  Week 16: number analyzed (Participants) | 51 | 26 | 26 | 7
  Week 16: No symptoms | 15 | 8 | 18 | 2
  Week 16: Mild | 14 | 6 | 6 | 4
  Week 16: Moderate | 15 | 7 | 2 | 1
  Week 16: Severe | 6 | 5 | 0 | 0
  Week 16: Very severe | 1 | 0 | 0 | 0

8. Secondary Outcome: Percentage Change From Baseline in Target and MRI-measurable Non- Target Lesion Volume in Group 1 and Group 2
Description: Percentage change from baseline in the sum of target lesion volume, MRI-measurable non-target lesion volume and all MRI measurable (target an non-target) lesion volume as assessed by BIRC.
  Target lesions are defined as anatomically reproducibly defined tissue(s) masses, which may be composed of one or several tissue types, and can be accurately measured by imaging technique MRI. Target lesion(s) (up to 3) should be identified at screening, be at least 2 cm in the longest diameter at baseline (for each selected lesion) and may be further reproducibly assessed by MRI.
  MRI-measurable non-target lesions are defined as all anatomic lesions other than selected as target and may be measured at radiologic assessment (at least 2 cm in the longest diameter at baseline, the volume may be further reproducibly assessed by MRI).
Time Frame: From Baseline up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2032-04

9. Secondary Outcome: Proportion of Participants With Changes From Baseline in Other Non-target Lesions in Group 1 and Group 2
Description: Percentage change from baseline in other non-target lesions (by BIRC). Non Target lesions are defined as:
  * Anatomic lesions, limb/trunkal areas affected by PROS, organomegaly when they may be measured only by caliper/ruler (e.g., circumference of changed limb or body part)
  * Truly non-measurable lesions (e.g., small lesions less than 2 cm on MRI, superficial visual lesions, masses, organomegaly, PROS-related enlargement of anatomic area identified by physical exam that is not measurable by reproducible imaging technique)
Time Frame: From Baseline up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2032-04

10. Secondary Outcome: Proportion of Participants With New Lesions in Group 1 and Group 2
Description: The proportion of patients with new lesions (as assessed by BIRC) will be assessed throughout the study.
Time Frame: From Baseline up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2032-04

11. Secondary Outcome: Pharmacokinetics (PK) of Alpelisib in Group 1 and Group 2: Maximum Concentration (Cmax)
Description: Maximum concentration of alpelisib following drug administration will be assessed for Group 1 and Group 2. After Week 28, blood samples will be collected only for participants who had dose escalation at next scheduled visit 4 weeks after the first dose escalation.
Time Frame: Week 17 Day 1 (Pre-dose, 1h post dose, 3h post dose, 5h post dose, 8h post dose , 24h post dose/ Pre-dose of Day 2), Week 20 Day 1 (Pre-dose, 3h post dose) and after Week 28, on Day 1 (Pre-dose and 3h post dose) 4 weeks after the first dose escalation
Reporting Status: Not Posted, anticipated posting 2032-04

12. Secondary Outcome: Pharmacokinetics (PK) of Alpelisib in Group 1 and Group 2: Trough Concentration (Ctrough)
Description: The trough observed concentration of alpelisib will be assessed for Group 1 and Group 2. After Week 28, blood samples will be collected only for participants who had dose escalation at next scheduled visit 4 weeks after the first dose escalation.
Time Frame: Week 17 Day 1 (Pre-dose and 24 h post dose/ Pre-dose of Day 2), Week 20 Day 1 (Pre-dose) and after Week 28, on Day 1 (Pre-dose) 4 weeks after the first dose escalation
Reporting Status: Not Posted, anticipated posting 2032-04

13. Secondary Outcome: Change From Baseline in Patient-reported Pain Assessed by Brief Pain Inventory (BPI) Worst Pain Intensity Item or Wong-Baker Faces Scale (Age Appropriate) in Pediatric and Adult Populations
Description: Change in scores from Brief Pain Inventory (BPI) items, or Wong-Baker Faces Scale (age appropriate). The BPI item that assesses worst pain intensity in the past 24 hours will be used to assess pain intensity for adult participants (≥18 years old) and pediatric participants (≥12 years old). Participants respond to the item on an 11-point numerical rating scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine). For children under 12, the Wong-Baker Faces Scale will be used in place of the BPI worst pain intensity item. This scale is a single-item that includes drawings of 6 faces that are associated with both a numeric rating and a descriptor (ranging from 0/no hurt - 10/hurts worst)
Time Frame: From Baseline up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2032-04

14. Secondary Outcome: Changes From Baseline in Patient-reported Health-related Quality of Life Assessed by PROMIS-profile (Patient Reported Outcome Measurement Information System) in Pediatric and Adult Populations
Description: Change in scores from the PROMIS-profile (Patient Reported Outcome Measurement Information System). The PROMIS Profiles are a group of PROMIS short forms measuring different domains of health-related quality of life (physical function, fatigue, ability to participate in social/peer relationships, pain interference, pain severity, anxiety, depression and sleep disturbance). All items include 5 response options, except for the pain intensity item, which has 11 response options.
Time Frame: From Baseline up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2032-04

15. Secondary Outcome: Changes From Baseline in Patient-reported Overall Impression of Symptoms Assessed by Patient Global Impression of Symptom Severity (PGIS) in Pediatric and Adult Populations
Description: Change in PGIS item. The PGIS is a single item to assess the participant's perception in the severity of their symptoms using a 5-point verbal rating scale, from "No symptoms" to "Very Severe".
Time Frame: From Baseline up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2032-04

16. Secondary Outcome: Duration of Response (DOR) in Participants Who Received Alpelisib in Group 1 and Group 2
Description: Duration of response (DOR) is defined as the time from first documented response until progression of PROS lesions by BIRC or death.
Time Frame: From first documented response until progression of PROS lesions or death, assessed up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2032-04

17. Secondary Outcome: Time to Treatment Failure in Participants Who Received Alpelisib in Group 1 and Group 2
Description: Time from randomization/alpelisib treatment start date until the discontinuation of study treatment due to lack of efficacy (including unsatisfactory therapeutic effect, disease progression) or safety reasons (including adverse events, death).
  Participants who complete the study or discontinue study treatment for other reasons (e.g. discontinuation due to Participant/Guardian decision, technical problems) will be censored at the date of last study treatment received.
Time Frame: From Baseline up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2032-04

18. Secondary Outcome: Overall Clinical Response Rate as Assessed by Investigator in Participants Who Received Alpelisib in Group 1 and Group 2
Description: Proportion of participants with overall clinical response reported as improvement, stable or worsening of clinical condition, as assessed by the investigator
Time Frame: Week 16, 24, 40, 48, 72, 96 and thereafter every 48 weeks
Reporting Status: Not Posted, anticipated posting 2032-04

19. Secondary Outcome: Proportion of Participants With Response During the Extension Period in Group 1 and Group 2
Description: Response (yes/no) at scheduled protocol visit. Response is defined by achieving at least 20% reduction from baseline in the sum of target lesion volumes (1 to 3 lesions, assessed by MRI by a blinded independent review committee (BIRC)), provided that none of the individual target lesions has ≥ 20% increase from baseline and in absence of progression of non-target lesions and without new lesions.
Time Frame: Week 40, 48, 72, 96, 144, 192, 240 and 264.
Reporting Status: Not Posted, anticipated posting 2032-04

20. Secondary Outcome: Changes in Symptoms and Complications/Comorbidities up to Week 16 on Treatment With Alpelisib as Compared to Placebo in Group 1 and Group 2
Description: Change in PROS-related symptoms and complications/comorbidities associated with PROS up to Week 16 among participants with symptoms and complications/comorbidities present at baseline
Time Frame: Baseline up to Week 16
Reporting Status: Not Posted, anticipated posting 2032-04

21. Secondary Outcome: Changes in Symptoms and Complications/Comorbidities Associated With PROS Over Time in Group 1 and Group 2
Description: Change in PROS-related symptoms and complications/comorbidities among participants with symptoms and complications/comorbidities present at baseline
Time Frame: Baseline up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2032-04

22. Secondary Outcome: Proportion of Participants With Healthcare Visit/Hospitalized Due to PROS in Group 1 and Group 2
Description: Proportion of participants with healthcare visit/hospitalized due to PROS will be assessed for Group 1 and Group 2.
Time Frame: From Baseline up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2032-04

23. Secondary Outcome: Proportion of Participants Requiring Rescue Surgery Due to PROS in Group 1 and Group 2
Description: Proportion of participants requiring rescue surgery due to PROS will be assessed for Group 1 and Group 2.
Time Frame: From Baseline up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2032-04

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to the cut-off date for the interim analysis (20-Mar-2024), approximately 35 months.
Description: The safety analysis were done on the safety population, which included all subjects who received at least one dose of study medication.
Groups:
- Group 1 (Greater or Equal to 18 Years) Alpelisib Period/Alpelisib Arm: Group 1 (Greater or equal to 18 years) Alpelisib period/Alpelisib arm: Events for participants initially randomized to Alpelisib who continued to active treatment after week 16 until primary analysis cut-off date.
- Group 1 (Greater or Equal to 18 Years) Alpelisib Period/Placebo Arm: Group 1 (Greater or equal to 18 years) Alpelisib period/Placebo arm: Events for participants initially randomized to Placebo who continued to active treatment after week 16 until primary analysis cut-off date.
- Group 1 (Greater or Equal to 18 Years) All Adults in Alpelisib Period: Group 1 (Greater or equal to 18 years) All adults in Alpelisib Period: All events for adults participants in the Alpelisib Period.
- Group 2 (6-17 Years) Alpelisib Period Alpelisib Arm: Group 2 (6-17 years) Alpelisib period Alpelisib arm: Events for participants initially randomized to Alpelisib who continued to active treatment after week 16 until primary analysis cut-off date.
- Group 2 (6-17 Years) Alpelisib Period Placebo Arm: Group 2 (6-17 years) Alpelisib period Placebo arm: Events for participants initially randomized to Placebo who continued to active treatment after week 16 until primary analysis cut-off date.
- Group 2 (6-17 Years) All Pediatrics in Alpelisib Period: Group 2 (6-17 years) All pediatrics in Alpelisib Period: All events for pediatrics participants aged 6-17 years old in the Alpelisib Period.
- Group 4 (2-5 Years) All Pediatrics: Group 4 (2-5 years) All pediatrics: All events for pediatrics participants aged 2-5 years old
- Group 5 (6-17 Years) All Pediatrics: Group 5 (6-17 years) All pediatrics: All events for pediatrics participants aged 6-17 years old.
Arm/Group | Group 1 (Greater or Equal to 18 Years) - Alpelisib Arm | Group 1 (Greater or Equal to 18 Years) - Placebo Arm | Group 1 (Greater or Equal to 18 Years) Alpelisib Period/Alpelisib Arm | Group 1 (Greater or Equal to 18 Years) Alpelisib Period/Placebo Arm | Group 1 (Greater or Equal to 18 Years) All Adults in Alpelisib Period | Group 2 (6-17 Years) - Alpelisib Arm | Group 2 (6-17 Years) - Placebo Arm | Group 2 (6-17 Years) Alpelisib Period Alpelisib Arm | Group 2 (6-17 Years) Alpelisib Period Placebo Arm | Group 2 (6-17 Years) All Pediatrics in Alpelisib Period | Group 4 (2-5 Years) All Pediatrics | Group 5 (6-17 Years) All Pediatrics
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/27 | 0/54 | 0/26 | 0/80 | 0/56 | 1/28 | 0/56 | 0/26 | 0/82 | 0/7 | 0/16
Serious Adverse Events (participants affected / at risk) | 5/54 | 2/27 | 16/54 | 3/26 | 19/80 | 3/56 | 2/28 | 8/56 | 2/26 | 10/82 | 3/7 | 2/16
Other Adverse Events (participants affected / at risk) | 47/54 | 24/27 | 52/54 | 26/26 | 78/80 | 45/56 | 21/28 | 53/56 | 23/26 | 76/82 | 7/7 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Greater or Equal to 18 Years) - Alpelisib Arm (N=54) | Group 1 (Greater or Equal to 18 Years) - Placebo Arm (N=27) | Group 1 (Greater or Equal to 18 Years) Alpelisib Period/Alpelisib Arm (N=54) | Group 1 (Greater or Equal to 18 Years) Alpelisib Period/Placebo Arm (N=26) | Group 1 (Greater or Equal to 18 Years) All Adults in Alpelisib Period (N=80) | Group 2 (6-17 Years) - Alpelisib Arm (N=56) | Group 2 (6-17 Years) - Placebo Arm (N=28) | Group 2 (6-17 Years) Alpelisib Period Alpelisib Arm (N=56) | Group 2 (6-17 Years) Alpelisib Period Placebo Arm (N=26) | Group 2 (6-17 Years) All Pediatrics in Alpelisib Period (N=82) | Group 4 (2-5 Years) All Pediatrics (N=7) | Group 5 (6-17 Years) All Pediatrics (N=16)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphatic malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb asymmetry (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adnexal torsion (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Greater or Equal to 18 Years) - Alpelisib Arm (N=54) | Group 1 (Greater or Equal to 18 Years) - Placebo Arm (N=27) | Group 1 (Greater or Equal to 18 Years) Alpelisib Period/Alpelisib Arm (N=54) | Group 1 (Greater or Equal to 18 Years) Alpelisib Period/Placebo Arm (N=26) | Group 1 (Greater or Equal to 18 Years) All Adults in Alpelisib Period (N=80) | Group 2 (6-17 Years) - Alpelisib Arm (N=56) | Group 2 (6-17 Years) - Placebo Arm (N=28) | Group 2 (6-17 Years) Alpelisib Period Alpelisib Arm (N=56) | Group 2 (6-17 Years) Alpelisib Period Placebo Arm (N=26) | Group 2 (6-17 Years) All Pediatrics in Alpelisib Period (N=82) | Group 4 (2-5 Years) All Pediatrics (N=7) | Group 5 (6-17 Years) All Pediatrics (N=16)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 3 | 0 | 3 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 9 | 1 | 13 | 3 | 16 | 5 | 2 | 14 | 7 | 21 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 2 | 2 | 4 | 3 | 1 | 7 | 2 | 9 | 1 | 1
Anal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 2 | 0 | 2 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 3 | 0 | 7 | 4 | 11 | 1 | 0 | 2 | 2 | 4 | 0 | 2
Defaecation disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 16 | 5 | 21 | 8 | 29 | 5 | 3 | 15 | 6 | 21 | 2 | 8
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 5 | 0 | 5 | 1 | 0 | 2 | 0 | 2 | 0 | 0
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 3 | 1 | 4 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 3 | 0 | 6 | 2 | 8 | 2 | 0 | 4 | 0 | 4 | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 4 | 8 | 1 | 9 | 5 | 2 | 8 | 3 | 11 | 1 | 1
Oral pain (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 5 | 0 | 5 | 2 | 0 | 3 | 0 | 3 | 0 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 3 | 3 | 0 | 6 | 2 | 8 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 4 | 2 | 6 | 6 | 2 | 10 | 7 | 17 | 4 | 5
Asthenia (General disorders) | 2 | 1 | 5 | 1 | 6 | 0 | 0 | 1 | 1 | 2 | 0 | 1
Chest pain (General disorders) | 1 | 3 | 3 | 0 | 3 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Fatigue (General disorders) | 2 | 4 | 3 | 5 | 8 | 5 | 3 | 8 | 1 | 9 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Haemorrhagic cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Induration (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inflammation (General disorders) | 1 | 0 | 6 | 1 | 7 | 1 | 0 | 4 | 2 | 6 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 4 | 1 | 5 | 0 | 0
Malaise (General disorders) | 1 | 0 | 4 | 0 | 4 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 3 | 0 | 1
Pyrexia (General disorders) | 5 | 0 | 8 | 2 | 10 | 5 | 1 | 17 | 8 | 25 | 4 | 5
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 4 | 1 | 5 | 0 | 1 | 1 | 0 | 1 | 1 | 0
COVID-19 (Infections and infestations) | 6 | 4 | 17 | 3 | 20 | 9 | 3 | 13 | 2 | 15 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 2 | 0 | 5 | 0 | 5 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dientamoeba infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 4 | 0 | 4 | 1 | 0
Fungal foot infection (Infections and infestations) | 1 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 7 | 1 | 8 | 1 | 1 | 3 | 2 | 5 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 3 | 1 | 1
Influenza (Infections and infestations) | 0 | 3 | 5 | 1 | 6 | 3 | 2 | 7 | 3 | 10 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 1 | 12 | 1 | 13 | 4 | 4 | 9 | 7 | 16 | 1 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 4 | 0 | 4 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 3 | 0 | 4 | 0 | 4 | 1 | 0 | 1 | 1 | 2 | 0 | 0
Sapovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scarlet fever (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 5 | 0 | 5 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 2 | 0 | 2 | 1 | 1 | 4 | 0 | 4 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 5 | 0 | 5 | 5 | 1 | 8 | 2 | 10 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 6 | 1 | 7 | 1 | 0 | 2 | 1 | 3 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 3 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 3 | 1 | 4 | 1 | 2
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Viral rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 1 | 4 | 0 | 0 | 1 | 1 | 2 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 3 | 1 | 0 | 1 | 1 | 2 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 4 | 2 | 6 | 1 | 0 | 3 | 1 | 4 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 4 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 5 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 2 | 2 | 5 | 2 | 7 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Lymph node palpable (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 4 | 0 | 5 | 3 | 8 | 1 | 0 | 3 | 1 | 4 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 1 | 6 | 4 | 10 | 4 | 1 | 6 | 1 | 7 | 2 | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 5 | 4 | 9 | 0 | 0 | 1 | 3 | 4 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 1 | 6 | 1 | 1 | 4 | 2 | 6 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 7 | 3 | 10 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Growth retardation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 10 | 3 | 13 | 2 | 1 | 13 | 4 | 17 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 4 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 10 | 4 | 16 | 6 | 22 | 11 | 3 | 20 | 5 | 25 | 2 | 2
Migraine (Nervous system disorders) | 1 | 1 | 3 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 1 | 2 | 3 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Encopresis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 2 | 0 | 2 | 1 | 0 | 3 | 0 | 3 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 2 | 0 | 3 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 8 | 0 | 8 | 4 | 1 | 7 | 2 | 9 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 5 | 0 | 5 | 6 | 0 | 9 | 2 | 11 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 3 | 0 | 3 | 0 | 3 | 1 | 0 | 2 | 0 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 1 | 21 | 4 | 25 | 1 | 0 | 6 | 2 | 8 | 1 | 3
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 2 | 6 | 6 | 12 | 1 | 0 | 1 | 1 | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 6 | 1 | 7 | 1 | 0 | 3 | 2 | 5 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 4 | 6 | 0 | 3 | 1 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 1 | 6 | 3 | 9 | 2 | 0 | 6 | 0 | 6 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT04589650/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT04589650/SAP_001.pdf